CLINICAL TRIAL: NCT02067039
Title: Evaluation of Rapid HIV Self-testing Among MSM in High Prevalence Cities
Brief Title: Evaluation of Rapid HIV Self-testing Among MSM (eSTAMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Emory University (Other); Northwestern University (Other); Public Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CDC-eSTAMP-41989
Record Dates: First submitted 2014-02-05; First posted 2014-02-20 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: HIV Infection
Keywords: HIV testing; Rapid HIV test; HIV self-testing; Men who have sex with men (MSM); HIV diagnosis; Sexual behavior
MeSH Terms: conditions — HIV Infections; Homosexuality; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV self-testing (Experimental): The intervention group of MSM (HIV negative or unaware of HIV status) will receive 4 rapid HIV test kits - 2 oral fluid tests (OraQuick), and 2 finger-stick blood tests (Sure Check). Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period, and men in the intervention arm will be allowed to order additional test kits to replenish the ones they use or give away. At month 12, all HIV-negative or those who are unaware of their HIV status participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a dried blood spot (DBS) specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing.
  Interventions: Device: OraQuick in home & Sure Check HIV tests
- Information only (No Intervention): All comparison group of MSM (HIV negative or unaware of HIV status) will take a baseline survey. Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period. At month 12, all HIV-negative and unaware of their HIV status comparison arm participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a DBS specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing.

INTERVENTIONS:
Device: OraQuick in home & Sure Check HIV tests — Provision of OraQuick in home & Sure Check HIV tests
  Arms: HIV self-testing

SUMMARY:
This study seeks to determine the public health impact of providing rapid HIV test kits to men who have sex with men (MSM) so they may test themselves at their convenience. The study will determine if men who receive the rapid HIV test kits report HIV testing at least three times per year. This study will be conducted in four consecutive parts. The first three parts are formative in nature to guide the development and implementation of Part 4 of the study. The research study will use two different types of rapid HIV tests. The OraQuick® In-Home HIV Test for oral fluid (FDA approved for home use) and Sure Check® HIV 1/2 Assay, currently FDA-approved for professional use and distributed in the U.S. as Clearview® Complete HIV-1/2 Rapid Test. An Investigational Device Exemption will be obtained from the FDA to allow the contractor to supply the Sure Check® HIV 1/2 Assay to study participants since it is not approved for home use.

DETAILED DESCRIPTION:
The eSTAMP project will evaluate the use and impact of providing rapid HIV tests for use to men who have sex with men (MSM) recruited via the internet. Data obtained through this study will include who will use the tests, how they were used, the utility of the tests in identifying HIV infections and promoting engagement in HIV care. This will inform policies to guide the optimal use of rapid HIV tests.

This research project will be conducted in four sequential parts to evaluate the acceptability, use and effectiveness of rapid HIV test kits among MSM in cities with high HIV prevalence. Each part will be independent and they will provide information to implement the next part of the study. At the end of each part, the data will be evaluated. The findings will guide the implementation of subsequent parts of the study.

Part 1 will evaluate the materials, packaging and instructions for conducting self-testing activities. MSM will be recruited from prior research studies or over the internet to participate in focus groups and in-depth interviews by Emory University or Northwestern University. These activities will take place in Atlanta, GA and Chicago, IL. Completed.

Part 2 will evaluate the user proficiency of participants performing the rapid HIV test on themselves while under observation using the instructional and materials developed in the previous part of the study. MSM who had participated in prior research studies and consented to future contact for involvement in additional studies were recruited by Emory University. Participants will conduct activities at Emory University in Atlanta, GA. Completed.

Part 3 will evaluate the performance of the rapid HIV tests by the proposed study population in real world settings. Participants will be recruited via the internet and directed to a research study site for further study activities. Participants will be shipped study materials (one OraQuick In-home HIV test, one SureCheck HIV 1/2 Assay and one dried blood spot (DBS) collection kit). Participants will report their rapid HIV test results online and return the DBS card for laboratory HIV testing. Completed.

Part 4 will evaluate the use and effectiveness of providing free rapid HIV tests as a public health strategy for increasing testing among MSM. We will recruit 3200 participants who report being HIV negative or unaware of their HIV status for the main trial. These participants will be randomly assigned to either the intervention or comparison condition after completing a baseline survey. An additional 150 MSM who report being HIV-positive will be recruited to evaluate the distribution of rapid HIV tests to their network partners.

Comparison arm: After completing the baseline survey, comparison arm participants will receive a welcome greeting and HIV prevention information. The online information will cover the importance of testing, links to AIDSVu and other resources to locate HIV testing services and prevention information in their area. Comparison arm participants will receive follow-up surveys at 3, 6, 9 and 12 months. After completing the 12 month assessment, participants will be sent a performance kit consisting of 1 oral fluid HIV test kit (OraQuick) and 1 finger-stick blood HIV test kit (Sure Check) and a DBS specimen collection kit that will be returned for HIV testing at the CDC laboratory.

Intervention arm: After completing the baseline survey, a welcome kit with 4 rapid HIV tests (2 oral fluid test kits [OraQuick] and 2 finger-stick blood test kits [Sure Check] will be sent to participants in the intervention arm to use and/or give away. Intervention arm participants will receive follow-up surveys at 3, 6, 9 and 12 months and have the option to order additional test kits at 3, 6 and 9 months to replenish kits that have been used or distributed. After completing the 12 month assessment, participants will be sent a performance kit consisting of 1 oral fluid HIV test kit (OraQuick) and 1 finger-stick blood HIV test kit (Sure Check) and a DBS specimen collection kit that will be returned for HIV testing at the CDC laboratory.

The men who report being HIV-positive who will be assigned to a one-arm descriptive cohort. Participants in this group will take a baseline survey and will receive rapid HIV test kits (OraQuick) to distribute to persons in their social and sexual networks (secondary users). Men in the HIV-positive group will complete a short follow-up survey at 3 months. Secondary users who use the tests will have access to study materials and referral information.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the Part 4 randomized controlled trial are:

  1. male sex at birth
  2. currently identify their sex as male
  3. able to provide informed consent
  4. at least 18 years of age
  5. report being HIV-negative or unaware of HIV status
  6. resident of United States and Puerto Rico.
  7. able to read instructions and complete study survey instruments in English
  8. reported anal sex with at least one man in the past 12 months
  9. have a valid email address, a cell phone capable of sending and receiving text messages, and a physical shipping address to receive kits
  10. never diagnosed with a bleeding disorder
  11. not part of an HIV vaccine trial
  12. not taking antiretroviral medication for HIV.

Exclusion Criteria:

* The exclusion criteria for the Part 4 randomized controlled trial are:

  1. not male sex at birth
  2. do not currently identify their sex as male
  3. not able to provide informed consent
  4. under 18 years of age
  5. report being HIV-positive
  6. not a resident of United States or Puerto Rico.
  7. not able to read instructions and complete study survey instruments in English
  8. do not report anal sex with at least one man in the past 12 months
  9. do not have a valid email address, a cell phone capable of sending and receiving text messages, or a physical shipping address to receive kits
  10. ever diagnosed with a bleeding disorder
  11. part of an HIV vaccine trial
  12. taking antiretroviral medication for HIV.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2665 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin MacGowan, MPH, Principal Investigator — Centers for Disease Control and Prevention; Pollyanna Chavez, PhD, Principal Investigator — Centers for Disease Control and Prevention; Patrick Sullivan, PhD, DVM, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Gwynn M, Chavez PR, Borkowf CB, Raiford JL, Gravens L, MacGowan RJ; eSTAMP Study Group. Pressure to Use HIV Self-Tests Among Men Who Have Sex With Men, United States, 2015-2016. AIDS Behav. 2022 Feb;26(2):623-630. doi: 10.1007/s10461-021-03422-6. Epub 2021 Aug 18. PMID 34406551
- [Derived] MacGowan RJ, Chavez PR, Borkowf CB, Owen SM, Purcell DW, Mermin JH, Sullivan PS; eSTAMP Study Group. Effect of Internet-Distributed HIV Self-tests on HIV Diagnosis and Behavioral Outcomes in Men Who Have Sex With Men: A Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):117-125. doi: 10.1001/jamainternmed.2019.5222. PMID 31738378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 3/2015 through 8/2015. Subjects were recruited online from internet (websites and music) catering to MSM.
Pre-assignment Details: Participants who did not provide contact information, complete and submit their baseline interview online, provided fraudulent information or later reported an HIV diagnoses before study enrollment were excluded.
Groups:
- Self-testing: The intervention group of MSM (HIV negative or unaware of HIV status) will receive 4 rapid HIV test kits - 2 oral fluid tests (OraQuick), and 2 finger-stick blood tests (Sure Check). Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period, and men in the intervention arm will be allowed to order additional test kits to replenish the ones they use or give away. At month 12, all HIV-negative or those who are unaware of their HIV status participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a dried blood spot (DBS) specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing. Participants had access to telephone consultation from study staff and a web-link to obtain HIV testing services in their community.
  OraQuick in home & Sure Check HIV tests: Provision of OraQuick in home & Sure Check HIV tests
- Control: All comparison group of MSM (HIV negative or unaware of HIV status) will take a baseline survey. Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period. At month 12, all HIV-negative and unaware of their HIV status comparison arm participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a DBS specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing. Participants had access to telephone consultation from study staff and a web-link to obtain HIV testing services in their community.
Period: Overall Study
Arm/Group | Self-testing | Control
Started | 1325 | 1340
3 Month Survey | 824 | 766
6 Month Survey | 735 | 756
9 Month Survey | 748 | 838
Completed (12 month survey) | 752 | 832
Not Completed | 573 | 508

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Self-testing | Information Only | Total
Number analyzed (Participants) | 1325 | 1340 | 2665
Age, Customized [Count of Participants; unit: Participants]
  Age-group: 18-29 years | 752 | 775 | 1527
  Age-group: >=30 years | 573 | 565 | 1138
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male Gender | 1325 | 1340 | 2665
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic white | 773 | 767 | 1540
  Race/ethnicity: Non-Hispanic black | 133 | 128 | 261
  Race/ethnicity: Hispanic | 296 | 324 | 620
  Race/ethnicity: Other/mixed | 123 | 121 | 244
Region of Enrollment [Number; unit: participants]
  United States | 1325 | 1340 | 2665
Recruitment site [Count of Participants; unit: Participants]
  Music | 510 | 553 | 1063
  Dating | 754 | 763 | 1517
  Social network | 61 | 24 | 85
HIV testing experience at enrollment [Count of Participants; unit: Participants]
  Never tested | 230 | 213 | 443
  Tested in past 12 months | 813 | 795 | 1608
  Tested more than 12 months ago | 282 | 332 | 614
At least 3 HIV tests in past year [Count of Participants; unit: Participants]
  Yes | 243 | 218 | 461
  No | 1082 | 1122 | 2204

OUTCOME MEASURES:

1. Primary Outcome: Frequency of HIV Testing by Internet-recruited MSM.
Description: Frequency of HIV testing >=3 times reported by participants over a 12-month follow-up period.
Time Frame: 12 months
Population: percent of MSM who reported testing at least three times over the course of the RCT
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing | Information Only
Number analyzed (Participants) | 1014 | 977
Participants | 777 | 215

2. Secondary Outcome: Linkage to HIV Testing and Care Services Following a Positive Rapid Test Result.
Description: MSM who report accessing supplemental testing and care following a positive rapid HIV test results.
Time Frame: 12 months
Population: Persons who reported initiating linkage to care following an HIV positive test
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing | Information Only
Number analyzed (Participants) | 25 | 11
Participants
  Linked to care | 16 | 10
  not linked to care | 9 | 1

3. Secondary Outcome: Newly Identified HIV Infections
Description: Report of positive HIV test result (self-test or provider testing)
Time Frame: 12 months
Population: All persons assigned to study.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing | Information Only
Number analyzed (Participants) | 1325 | 1340
Participants | 25 | 11

4. Secondary Outcome: HIV Infections Among Social Network Associates
Description: Number of social network associates (N=2150)who received a study self-test from ST participants (N=1325) and who reported a positive HIV self-test result. Sample size for this analyses is 2150.
Time Frame: 12 months
Population: Number of social network associates who used a study HIV self-test and received a new HIV diagnosis
Measure: Number; unit: social network members
Groups:
- Self-testing Social Network Associates (N=2150): The intervention group of MSM (HIV negative or unaware of HIV status) will receive 4 rapid HIV test kits - 2 oral fluid tests (OraQuick), and 2 finger-stick blood tests (Sure Check). Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period, and men in the intervention arm will be allowed to order additional test kits to replenish the ones they use or give away. At month 12, all HIV-negative or those who are unaware of their HIV status participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a dried blood spot (DBS) specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing. Participants had access to telephone consultation from study staff and a web-link to obtain HIV testing services in their community.
  OraQuick in home & Sure Check HIV tests: Provision of OraQuick in home & Sure Check HIV tests
- Control: Control group did not distribute HIV self-tests to social network members
Arm/Group | Self-testing Social Network Associates (N=2150) | Control
Number analyzed (Participants) | 2150 | 0
social network members | 34 |

ADVERSE EVENTS:
Time Frame: From initiation of study enrollment though final reporting of study data: 20 months.
Description: Participants could call to study phone number or report events via email to study staff or Emory University IRB.
Groups:
- OraQuick in Home & Sure Check HIV Tests: The intervention group of MSM (HIV negative or unaware of HIV status) will receive 4 rapid HIV test kits - 2 oral fluid tests (OraQuick), and 2 finger-stick blood tests (Sure Check). Men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 12-month follow-up period, and men in the intervention arm will be allowed to order additional test kits to replenish the ones they use or give away. At month 12, all HIV-negative or those who are unaware of their HIV status participants will be sent 1 oral fluid test (OraQuick), 1 finger-stick blood test (Sure Check), and a dried blood spot (DBS) specimen collection kit to be mailed to Emory University after collecting a blood sample for laboratory testing.
  OraQuick in home & Sure Check HIV tests: Provision of OraQuick in home & Sure Check HIV tests
Arm/Group | OraQuick in Home & Sure Check HIV Tests | Information Only
All-Cause Mortality (participants affected / at risk) | 0/1325 | 0/1340
Serious Adverse Events (participants affected / at risk) | 0/1325 | 0/1340
Other Adverse Events (participants affected / at risk) | 0/1325 | 0/1340

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes